CLINICAL TRIAL: NCT05316961
Title: Clinical Effectiveness of Pulsed Electromagnetic Field Therapy as a Treatment Adjunct to Eccentric Exercise for Achilles Tendinopathy: a Randomized Controlled Trial
Brief Title: Clinical Effectiveness of PEMF as a Treatment Adjunct to Eccentric Exercise for Achilles Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Assistant Professor (Clinical) of Orthopaedics & Traumatology, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021.150-T
Record Dates: First submitted 2022-01-12; First posted 2022-04-07 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Achilles Tendinopathy
Keywords: Pulsed electromagnetic field therapy; Eccentric exercise; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEMF group (Experimental): Participants will receive active pulsed electromagnetic field therapy two times a week for eight weeks. The options of the appliance will be adjusted to 1.5 mT, 10Hz on one leg for 10 minutes. A total of 16 sessions will be given to each participant. Each session will last for 10 minutes. Participants will be positioned in sitting on a chair comfortably. They will receive intervention at Prince of Wales hospital.
  3 sets of 10 repetitions of the eccentric exercises are carried out once daily for 6 weeks and after 6 weeks, the patients are instructed to carry out 3 sets of 10 repetitions, 3 times per week for 6 more weeks. The intensity of the exercise should be such that pain, or discomfort, is experienced in the last set of 10 repetitions.
  Interventions: Device: Active PEMF; Other: Eccentric exercise
- Sham group (Sham Comparator): Participants will receive sham pulsed electromagnetic field therapy two times a week for eight weeks. The options of the appliance will be adjusted to 0 mT, 0Hz on one leg for 10 minutes. A total of 16 sessions will be given to each participant. Each session will last for 10 minutes. Participants will be positioned in sitting on a chair comfortably. They will receive intervention at Prince of Wales hospital.
  3 sets of 10 repetitions of the eccentric exercises are carried out once daily for 6 weeks and after 6 weeks, the patients are instructed to carry out 3 sets of 10 repetitions, 3 times per week for 6 more weeks. The intensity of the exercise should be such that pain, or discomfort, is experienced in the last set of 10 repetitions.
  Interventions: Device: Sham PEMF; Other: Eccentric exercise

INTERVENTIONS:
Device: Active PEMF — PEMF 1.5mT, 10Hz, 10 minutes
  Arms: PEMF group
Device: Sham PEMF — PEMF 0mT, 0Hz, 10 minutes
  Arms: Sham group
Other: Eccentric exercise — Eccentric exercise, 10 repetitions, 3 sets

SUMMARY:
This study aims to investigate the clinical effectiveness of PEMF as an adjunct to a program of eccentric exercise for the treatment of Achilles tendinopathy. The study objective is to establish whether PEMF plus eccentric exercise in people with Achilles tendinopathy will improve rehabilitation outcomes compared to eccentric exercise only. This study also investigates the effects of PEMF on pain, functional outcomes, mechanical and morphological properties of tendon among patients with Achilles tendinopathy. Investigators hypothesize that pulsed electromagnetic field therapy is effective in reducing pain, improving functional outcomes, and restoring mechanical and morphological properties of tendons in patients with Achilles tendinopathy.

This study is a double-blinded, randomized controlled trial to investigate the clinical effects of pulsed electromagnetic field therapy (PEMF) for Achilles tendinopathy. Participants will be recruited from the outpatient clinic of the orthopedic and traumatology department at Prince of Wales Hospital. Fifty-four patients aged between 18 and 70 with Achilles tendinopathy will be invited to join this trial after informed consent. Participants will be randomized to any of the 2 groups: the intervention group (n=27; PEMF (Quantum Tx) treatment), and the control group (n=27; sham treatment with dummy exposure to PEMF).

Baseline measurements of all self-reported outcomes, functional outcomes, and ultrasound imaging assessments, such as ankle range of motion, jumping ability, pain level, calf muscle strength, calf muscle endurance, physical activity level, quality of life by SF-36 will be measured.

DETAILED DESCRIPTION:
Randomization and blinding Participants will be randomized into 1:1 allocation, blocked randomization with 27 participants in the PEMF group and 27 participants in the sham group. Each allocation will be assigned with a unique RFID (generated during block randomization by the PEMF supplier service) recognizable by the PEMF machine. The participants will be assigned an RFID by which the PEMF or sham treatment will be randomly assigned to the RFID. A biostatistician who does not participate in the recruitment of patients will oversee the randomization. Hence, both participants and the research personnel are blinded, and participants will use the RFID to complete the assigned treatment without knowing which treatment they are receiving.

Intervention The intervention will be held at the Chinese University of Hong Kong. Participants in the intervention group will be exposed to PEMF treatment by a PEMF device (Quantum Tx, Singapore). The active PEMF device does not produce heat or cause any sensation to the tissue which allows the participants to be blinded to the treatment. Participants in the control group will receive a sham exposure with the same PEMF device. The diseased leg will be exposed to PEMF or sham treatment for 10 minutes per session, and the treatment regime will run twice a week for 8 weeks, summing up 16 sessions of PEMF or sham exposure in total.

The procedure of PEMF treatment is shown as follows:

The subject will be seated at a 90 degrees position on a chair. The solenoids of the PEMF device will be adjusted to be over the foot and ankle (Achilles tendon and lower calf muscle).

The options of the appliance will be adjusted to 1.5mT, 10Hz on the diseased leg for 10 minutes.

In addition to PEMF, all participants will also perform eccentric calf muscle exercise. The first step is stretching exercises for the calf muscles. The stretching is a static stretch of the gastrocnemius (knee in extension) and soleus (knee in flexion). The participants are instructed to hold these at least for 30s and repeat each exercise three times. There is a 1-min rest between each stretch. 3 sets of 10 repetitions of the eccentric exercises are carried out once daily for 6 weeks and after 6 weeks, the participants are instructed to carry out 3 sets of 10 repetitions, 3 times per week for 6 more weeks. The intensity of the exercise should be such that pain, or discomfort, is experienced in the last set of 10 repetitions. Every session ended with the same static stretch exercise as in step 1. If a participant is unable to complete 3 sets of 15 repetitions, the participant is instructed to start with a lower number of repetitions and/or sets (a minimum of 2 sets of 10) and progress to the full amount as able.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70
* Tenderness with palpation 2-6 cm above the Achilles tendon insertion on the calcaneus (midportion Achilles tendinopathy)
* Recurrent complaints in 1 or both Achilles' tendons at rest and/or during exercise for the preceding 3 month
* Structural changes of the tendon were confirmed via sonographic examination during the initial physical exam
* Achilles tendinopathy affecting the insertional and mid-portion of the Achilles tendon
* Clinical symptoms associated with Achilles tendinopathy that do not respond well to conventional conservative treatments before entering the study
* Informed consent

Exclusion Criteria:

* History of surgery on the affected lower limb in the past year
* Mental/physical limitation rendering participant to follow instructions
* With medical or musculoskeletal problems that could affect the ability to complete assessments (i.e. with walking aids or wheel-chaired)
* Severe cognitive impairments and neurological disorders that will affect data collection by questionnaires
* Fractures of the trained body parts within the past 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from baseline to 6 months
  The Visual Analogue Scale (VAS) requires participants to rate their pain on a defined scale from 0-10. 0 refers to no pain while 10 refers to severe pain. Lower scores mean a better outcome.
Victorian Institute of Sport Assessment - Achilles questionnaire (VISA-A) | Change from baseline to 6 months
  The Victorian Institute of Sport Assessment - Achilles questionnaire (VISA-A) is used to evaluate the clinical severity of patients, monitor the change in symptoms and function following interventions provided for Achilles tendinopathy. The questionnaire contains eight questions, covering three necessary domains: 1) pain, 2) functional status, and 3) activity. The first seven questions have a score out of 10, and question 8 scores a maximum of 30. The minimum value is 0 and the maximum value is 100. Higher scores mean a better outcome. Asymptomatic individuals may score 100 points in VISA-A.

SECONDARY OUTCOMES:
Ankle range of motion | Change from baseline to 6 months
  A standard goniometer will be used to measure the range of motion (ROM) of ankle dorsiflexion. It will be used as an indicator of the flexibility of the gastrocnemius muscle. The participant will maximally dorsiflex the ankle while keeping the knee extended and the heel on the floor.
Calf muscle endurance | Change from baseline to 6 months
  The heel-rise test will be used to measure calf-muscle endurance. The participant will start from standing on a pressure mat (Tekscan, U.S.). The information on the plantar pressure will be collected for analyses. The participant will be instructed to rise as high as possible on the heel each time until fatigue. The participant should keep the knees straight. The participant can place 2 fingertips per hand on the wall to maintain balance. The rhythm will be set at a frequency of 30 heel rises per minute by following a metronome. The number of repetitions, maximum heel-rise height, and the total amount of work performed are recorded.
Tendon thickness | Change from baseline to 6 months
  The thickness (mm) of each tendon were measured with axial (i.e., perpendicular to the direction of the fibers) grayscale ultrasound 2 cm and 3 cm from the end of the tendon.
Neovascularity | Change from baseline to 6 months
  The Achilles tendons were examined in longitudinal plane. The location and number of neovessels observed with Power Doppler Ultrasound were scored using the modified Öhberg score.6,14 This score was recorded as 0 (no vessels visible), 1+ (1 vessel, mostly anterior to the tendon), 2+ (1 or 2 vessels throughout the tendon), 3+ (3 vessels throughout the tendon), or 4+ (more than 3 vessels throughout the tendon).
Tendon elasticity | Change from baseline to 6 months
  The mechanical properties of tendons will be measured by Shear-wave elastography (SWE) performed using an Aixplorer (Supersonic Imagine, Aix-en-Provence, France), a form of ultrasound imaging. It can detect changes in mechanical properties that are associated with tendon healing that is closely correlated with symptoms. The participant will be positioned in prone lying with feet hanging over the plinth to allow ankle movement during the sonographic exam. The resting ankle range of motion is measured by a goniometer.
Short Form 36 questionnaire (SF-36) | Change from baseline to 6 months
  Short Form 36 questionnaire (SF-36) will be used to evaluate health-related quality of life. SF-36 covers a variety of domains, including bodily pain, physical function, mental health, and social health of the participants. The minimum value is 0 and the maximum value is 100. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ka-Kin Samuel Ling, MSc, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- KO Man Chi, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Ko VM, Chen SC, He X, Fu SC, Franco-Obregon A, Yung PS, Ling SK. Short-term Effects of Pulsed Electromagnetic Field Therapy for Achilles Tendinopathy: A Randomized Controlled Trial. Orthop J Sports Med. 2024 Nov 12;12(11):23259671241284772. doi: 10.1177/23259671241284772. eCollection 2024 Nov. PMID 39534390
- [Derived] Ko VM, He X, Fu SC, Yung PS, Ling SK. Clinical effectiveness of pulsed electromagnetic field therapy as an adjunct treatment to eccentric exercise for Achilles tendinopathy: a randomised controlled trial. Trials. 2023 Jun 12;24(1):394. doi: 10.1186/s13063-023-07434-6. PMID 37308969